CLINICAL TRIAL: NCT03615001
Title: Assessing the Performance, Safety and Usability of Our Next Generation T-DOC® NXT Catheter for Performing Urodynamic Studies
Brief Title: T-DOC® NXT Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TDOC-NXT-01
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Incontinence, Urge
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Urodynamics Arm (Experimental)
  Interventions: Device: TDOC NXT

INTERVENTIONS:
Device: TDOC NXT — Assessing the Performance, Safety and Usability of our Next Generation T-DOC® NXT Catheter for Performing Urodynamic Studies

SUMMARY:
Assessing the Performance, Safety and Usability of our Next Generation T-DOC® NXT Catheter for Performing Urodynamic Studies

ELIGIBILITY:
Inclusion Criteria:

* Male and Female (Adult age 21+)
* Patients with clinical indication for urodynamics (UDS) testing, for any medically necessary reason as per the physician.

Exclusion Criteria:

* Patients who suffer from bladder infections (not including patients with asymptomatic bacteriuria)
* Patients who are pregnant
* Patients with recent (less than 2 weeks) pelvic floor surgery
* Patients who require the use of a suprapubic catheter
* Patients with significant cognitive deficiency that prevent the patient from giving informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Franklin Square Hospital/White Marsh, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Urodynamics Arm: Urodynamic testing and data collection (per protocol) using the TDOC NXT catheters
Period: Overall Study
Arm/Group | Urodynamics Arm
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Urodynamics Arm
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients in Which the T-DOC® NXT Catheters Are Safe in Measuring Urodynamic Pressure in Adults.
Description: A binary clinician response after each UDS study is used to assess if it is clinically adequate (success) or inadequate (failure) in each patients questionnaire and presented to the clinician where safety (Yes the device is safe and No the device is not safe) will be reported. A minimum of 20 patient questionnaires is required to answer "YES" the device is safe for a positive outcome and a maximum of 40.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Urodynamics Arm
Number analyzed (Participants) | 20
Participants | 20

2. Primary Outcome: The Number of Patients in Which the T-DOC® NXT Catheters Are Effective in Measuring Urodynamic Pressure in Adults.
Description: A binary clinician response after each UDS study is used to assess if it is clinically adequate (success) or inadequate (failure) in each patients questionnaire and presented to the clinician where effectiveness (Yes the device is effective and No the device is not effective) will be reported. A minimum of 20 patient questionnaires is required to answer "YES" the device is effective for a positive outcome and a maximum of 40.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Urodynamics Arm
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: Through study completion (average of one day)
Arm/Group | Urodynamics Arm
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT03615001/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT03615001/SAP_001.pdf